CLINICAL TRIAL: NCT00948805
Title: Evaluation of the Luteolytic Effect of a Gonadotropin Releasing Hormone (GnRH) Agonist After the Administration of Human Chorionic Gonadotropin (hCG) in the Initial Follicular Phase a Its Influence on the Prognosis of in Vitro Fertilization Treatment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Cláudia Messias Gomes, Gynecology of Faculty of Medicine of the University of SãoPaulo (Disciplina de Ginecologia da Faculdade de Medicina da Universidade de São Paulo)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0555/09
Record Dates: First submitted 2009-07-23; First posted 2009-07-29 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: Infertility
Keywords: corpus luteum rescue; Gonadotropin Releasing Hormone (GnRH agonist); human Chorionic Gonadotropin (hCG); infertility; pregnancy rate
MeSH Terms: conditions — Infertility | interventions — Gonadotropin-Releasing Hormone; Ovidrel; Goserelin; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GnRH agonist (Experimental): 3,6 mg of goserelin acetate (GnRH agonist) will be administered on the 21st day of the menstrual cycle previous to ovarian stimulation. 250 mg of hCG will be administered on the first day of menses and a starting dose of 150 IU of FSH will be started 2 days later as a part of a long ovarian stimulation protocol. Ovulation will be triggered with a 250 mg of hCG when at least 2 follicles attain 18mm and to accommodate oocyte retrieval within 36 hours.
  Interventions: Drug: GnRH agonist
- Control (Active Comparator): 250 mg of hCG will be administered on the first day of menses and a starting dose of 150 IU of FSH will be started 2 days later as a part of a long ovarian stimulation protocol. Ovulation will be triggered with a 250 mg of hCG when at least 2 follicles attain 18mm and to accommodate oocyte retrieval within 36 hours.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: GnRH agonist — 3,6mg of goserelin acetate, 250mg of hCG, FSH variable dose according to the number of days required for appropriate ovarian stimulation
  Other Names: Ovidrel; Zoladex; Gonal
  Arms: GnRH agonist
Drug: Control — 250mg of hCG, Zoladex, FSH variable dose according to the number of days required for appropriate ovarian stimulation
  Other Names: Zoladex; Ovidrel; Gonal
  Arms: Control

SUMMARY:
This study was designed to evaluate the ability of gonadotropin releasing hormone (GnRh) agonist to prevent the rise of progesterone during controlled ovarian stimulation for in vitro fertilization (IVF) after the administration of human Chorionic Gonadotropin (hCG) on the first day of menses.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of a GnRH agonist in preventing the functional rescue of corpus luteum in women submitted to controlled ovarian stimulation with administration of hCG on the first day of menses and to evaluate its effect on pregnancy rate and ovarian steroidogenesis.

ELIGIBILITY:
Inclusion Criteria:

* age >21 and < 38 years old
* polycystic ovarian syndrome
* risk for ovarian hyperstimulation syndrome

Exclusion Criteria:

* recurrent abortion
* endometriosis
* more than 3 IVF failures
* use of oral contraceptive pills in the preceding 3 months
* low response to gonadotropins

Ages: 21 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Frequency of functional rescue of corpus luteum | 6 months

SECONDARY OUTCOMES:
Pregnancy rate | 6 months
Levels of serum steroids | 6 months
Levels of serum gonadotropins | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Serafini, PhD, Study Chair — Gynecology of Faculty of Medicine of University of SãoPaulo (Disciplina de Ginecologia da Faculdade de Medicina da Universidade de São Paulo)
Locations (1):
- Assisted Reproduction Center "Governor Mário Covas" of the Faculty of Medicine of the University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: University of São Paulo web page — http://www.fm.usp.br